CLINICAL TRIAL: NCT03993912
Title: A Phase III Study Comparing Lenalidomide and Subcutaneous Daratumumab (R-Dara SC) vs Lenalidomide and Dexamethasone (Rd) in Frail Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High Dose Therapy
Brief Title: Compare Lenalidomide and Subcutaneous Daratumumab vs Lenalidomide and Dexamethasone in Frail Subjects With Previously Untreated Multiple Myeloma Who Are Ineligible for High Dose Therapy
Acronym: IFM2017_03
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018_16; 2018-003535-30 (EudraCT Number)
Record Dates: First submitted 2019-05-27; First posted 2019-06-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Newly diagnosed Multiple Myeloma; Frail elderly patients; Dexamethasone-sparing regimen; Daratumumab; Toxicity
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Experimental group (Experimental): Daratumumab SC 1800 mg
  * once every week for 8 weeks
  * then once every other week for 16 weeks
  * thereafter once every 4 weeks, until progression Lenalidomide PO (25mg): days 1 through 21 of each 28-day cycle, until progression Dexamethasone PO (20mg): days 1, 8, 15, 22 of a 28-day cycle, for the first 2 cycles, then discontinued
  Interventions: Drug: Daratumumab SC in combination with Lenalidomide; Drug: Lenalidomide PO (25mg); Drug: Dexamethasone PO (20mg): days 1, 8, 15, 22 of each 28-day cycle, until progression
- Arm 2: Control group (Sham Comparator): Lenalidomide PO (25mg): days 1 through 21 of each 28-day cycle, until progression Dexamethasone PO (20mg): days 1, 8, 15, 22 of each 28-day cycle, until progression
  Interventions: Drug: Lenalidomide PO (25mg); Drug: Dexamethasone PO (20mg): days 1, 8, 15, 22 of each 28-day cycle, until progression

INTERVENTIONS:
Drug: Daratumumab SC in combination with Lenalidomide — Daratumumab SC 1800 mg
  * once every week for 8 weeks
  * then once every other week for 16 weeks
  * thereafter once every 4 weeks, until progression
  Arms: Arm 1: Experimental group
Drug: Lenalidomide PO (25mg) — Lenalidomide PO (25mg): days 1 through 21 of each 28-day cycle, until progression
Drug: Dexamethasone PO (20mg): days 1, 8, 15, 22 of each 28-day cycle, until progression — Dexamethasone PO (20mg): days 1, 8, 15, 22 of each 28-day cycle, until progression

SUMMARY:
This is a Phase 3, randomized (study drug assigned by chance), open-label (participants and researchers are aware about the treatment, participants are receiving), active-controlled (study in which the experimental treatment or procedure is compared to a standard treatment or procedure), parallel-group (each group of participants will be treated at the same time), and multicenter (when more than one hospital team work on a medical research study) study in participants with newly diagnosed multiple myeloma (a blood cancer of plasma cells) and who are not candidates for high dose chemotherapy (treatment of disease, usually cancer, by chemical agents) and autologous stem cell transplant (ASCT). The primary hypothesis of this study is that subcutaneous Daratumumab in combination with Lenalidomide will prolong progression-free survival and likely induce less toxicity as compared with Lenalidomide and dexamethasone, in elderly frail subjects with newly diagnosed Multiple myeloma who are ineligible for high dose chemotherapy and ASCT

DETAILED DESCRIPTION:
The primary hypothesis of this study is that subcutaneous Daratumumab in combination with Lenalidomide will prolong progression-free survival and likely induce less toxicity as compared with Lenalidomide and dexamethasone, in elderly frail subjects with newly diagnosed Multiple myeloma who are ineligible for high dose chemotherapy and ASCT

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 65 years of age.
2. Subject must have documented multiple myeloma satisfying the CRAB criteria and measurable disease.
3. Newly diagnosed and not considered candidate for high-dose chemotherapy with SCT.
4. Subject must have a Frailty Score ≥ 2
5. Subject must have within 5 days prior to first drug intake (C1D1) pretreatment clinical laboratory values meeting the following criteria during the Screening Phase:

   * hemoglobin ≥7.5 g/dL
   * absolute neutrophil count ≥1.0 x 109/L
   * platelet count ≥70 x 109/L
   * aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN)
   * alanine aminotransferase (ALT) ≤2.5 x ULN
   * total bilirubin ≤2.0 x ULN
   * creatinine clearance≥30mL/min
6. Measurable ISS with β2-microglobulin and albumin values for randomization
7. A man who is sexually active with a woman of childbearing potential must agree to use a latex or synthetic condom, even if they had a successful vasectomy. All men must also not donate sperm during the study, for 4 weeks after the last dose of lenalidomide, and for 4 months after the last dose of daratumumab. Women participating in this study must be postmenopausal.
8. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.
9. Subjects affiliated with an appropriate social security system.

Exclusion Criteria:

1. Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma.
2. Subject has a diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
3. Subject has prior or current systemic therapy or SCT for multiple myeloma
4. Subject has a history of malignancy (other than multiple myeloma) within 5 years before the date of randomization
5. Subject has had radiation therapy within 14 days of randomization.
6. Subject has had plasmapheresis within 28 days of randomization.
7. Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
8. Subject has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume [FEV] in 1 second <60% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (intermittent asthma is allowed).
9. Subject is known to be seropositive for history of human immunodeficiency virus (HIV)
10. Seropositive for hepatitis B.
11. (Known to be) seropositive for hepatitis C
12. Subject has any concurrent medical or psychiatric condition or disease that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
13. Subject has clinically significant cardiac disease, including:

    * myocardial infarction within 1 year before randomization, or an unstable or uncontrolled disease/condition related to or affecting cardiac function
    * uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities
    * screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec
14. Subject has known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients
15. Subject has plasma cell leukemia or POEMS syndrome
16. Subject is known or suspected of not being able to comply with the study protocol. Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject or that could prevent, limit, or confound the protocol-specified assessments.
17. Subject has had major surgery within 2 weeks before randomization or has not fully recovered from surgery.
18. Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before randomization or is currently enrolled in an interventional investigational study.
19. Refusal to consent or protected by legal regime ( guardianship, trusteeship)
20. Subject has contraindications to required prophylaxis for deep vein thrombosis and pulmonary embolism
21. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 294 (Estimated)
Dates: Start 2019-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Comparison of the efficacy of Daratumumab SC injection when combined with Lenalidomide (R-Dara SC) vs Lenalidomide and Dexamethasone (Rd): PFS | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  The primary objective is to compare the efficacy of Daratumumab SC injection when combined with Lenalidomide (R-Dara SC) to that of Lenalidomide and Dexamethasone (Rd), in terms of PFS in frail subjects with newly diagnosed myeloma who are not candidates for high dose chemotherapy and autologous stem cell transplant.

SECONDARY OUTCOMES:
Time-to-treatment failure | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
Time-to-next treatment | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
PFS2 time | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
Overall survival (OS) time | From date of randomization until the date of death from any cause, whichever came first, assessed up to 84months
  Overall survival (OS) time,
Complete remission (CR) | From date of randomization until the date of first documented progression whichever came first, assessed up to 84months
  Percentage of participants with CR, as defined by the IMWG criteria, will be reported.
Very good partial response (VGPR) or better. | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  VGPR or better, defined as VGPR or CR according to the IMWG criteria during or after the study treatment at the time of data cutoff.
Overall response (CR + VGPR + partial response [PR]). | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Overall response, defined as CR or VGPR or PR, according to the IMWG criteria
Occurrence of grade 3 or more side effects. | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Collecting all AE (grade 3 or more)
Safety and tolerability of Daratumumab SC when administered in combination with Revlimid: NCI-CTCAE V5.0. | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Evaluation of safety data by type, frequency, severity, relation to study drug, according to NCI-CTCAE V5.0.
Evaluation of quality of life based on MY20 questionnaires | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Treatment effects on patient reported outcomes and heath economic/resource utilization.
Evaluation of quality of life based on EORTC C30 questionnaires | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Treatment effects on patient reported outcomes and heath economic/resource utilization.
Evaluation of quality of life based on EQ-5D questionnaires | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months
  Treatment effects on patient reported outcomes and heath economic/resource utilization.
Minimal residual disease (MRD) negative rate at 12 months. | after 12 months of treatment
  Proportion of participants assessed as MRD negative
Event Free Survival | From date of randomization until the date of first documented progression or date of toxicity or date of death from any cause, whichever came first, assessed up to 84months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Facon, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (23):
- France (23):
  - Chru Jean Minjoz, Besançon
  - Ch Blois Simone Veil, Blois
  - Ch Fleyriat, Bourg-en-Bresse
  - Chru Brest Site Hopital Morvan, Brest
  - Chu de Caen Normandie, Caen
  - Hopital Prive Sevigne - Cesson, Cesson-Sévigné
  - Chu Dijon Bourgogne, Dijon
  - Chu de Grenoble, Grenoble
  - Gpe Hospitalier La Rochelle-Re-Aunis, La Rochelle
  - Ch Chartres Louis Pasteur-Le Coudray, Le Coudray
  - Hôpital Claude Huriez, CHU, Lille
  - Institut Paoli Calmettes, Marseille
  - Chi Mont de Marsan Et Pays Des Sources, Mont-de-Marsan
  - Chu Montpellier, Montpellier
  - Chu de Nantes Site Hotel Dieu Hme, Nantes
  - Chu de Nice Hopital de L'Archet, Nice
  - Hopital Haut-Leveque - Chu, Pessac
  - Centre Hospitalier de Perigueux, Périgueux
  - Chru Rennes Site Pontchaillou, Rennes
  - Centre Hospitalier de Saint Quentin, Saint-Quentin
  - Centre Hospitalier Saint-Malo, St-Malo
  - Oncopole Chu Toulouse, Toulouse
  - Chu de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Manier S, Lambert J, Hulin C, Macro M, Laribi K, Araujo C, Pica GM, Touzeau C, Godmer P, Slama B, Karlin L, Orsini Piocelle F, Dib M, Sanhes L, Morel P, El Yamani A, Tiab M, Tabrizi R, Richez V, Garderet L, Royer B, Bareau B, Mariette C, Fleck E, Robu D, Calmettes C, Rigaudeau S, Demarquette H, Frenzel L, Decaux O, Mohty M, Arnulf B, Bigot N, Perrot A, Corre J, Mary JY, Avet-Loiseau H, Moreau P, Leleu X, Facon T. Safety and efficacy of a dexamethasone-sparing regimen with daratumumab and lenalidomide in patients with frailty and newly diagnosed multiple myeloma (IFM2017-03): a phase 3, open-label, multicentre, randomised, controlled trial. Lancet Oncol. 2025 Oct;26(10):1323-1333. doi: 10.1016/S1470-2045(25)00280-3. PMID 41038184